CLINICAL TRIAL: NCT02540187
Title: Tissue Factor Pathway Inhibitor (TFPI) and Haemorrhagic Manifestations in Haemophilia A and B Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 1108164
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Hemophilia
Keywords: haemophilia; TFPI; thrombin generation; hemorrhagic score
MeSH Terms: conditions — Hemophilia A | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood specimen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- haemophilia A: 1. Blood specimen for measuring :
     * Free TFPI and TFPI activity levels
     * Thrombin generation in platelet rich plasma (PRP) and platelet poor plasma (PPP)
     * Thrombin generation assay (TGA) in fresh PRP and frozen PPP
  2. Hemorrhage score for each patient
  Interventions: Other: blood specimen
- Haemophilia B: 1. Blood specimen for measuring :
     * Free TFPI and TFPI activity levels
     * Thrombin generation in platelet rich plasma (PRP) and platelet poor plasma (PPP)
     * Thrombin generation assay (TGA) in fresh PRP and frozen PPP
  2. Hemorrhage score for each patient
  Interventions: Other: blood specimen

INTERVENTIONS:
Other: blood specimen

SUMMARY:
Haemophilia is a rare and serious congenital defect of blood coagulation due to a genetic mutation on a sexual chromosome. It affects quasi-essentially the men and it is responsible for bleeding. There are two types of haemophilia: Haemophilia A, (85 % of cases), due to a factor VIII (FVIII) deficiency and Haemophilia B (15 % of cases) due to factor IX (FIX) deficiency. According to the intensity of the defect, there are three forms of haemophilia: severe (FVIII or FIX lower than 1 %), moderate (factor level between 1 and 5 %), minor (factor level between 5 and 40 %). For a same level of factor VIII or IX, hemorrhagic manifestations are variable from one patient to the other. Moreover, several studies showed that haemophilic B patients bleed less and consume fewer anti-hemophilic concentrate that haemophilic A patients.

The main inhibitors of the coagulation are antithrombin, Protein C-Protein S-Thrombomodulin system, and tissue factor pathway inhibitor (TFPI). TFPI is the specific and exclusive inhibitor of tissue factor pathway that is the main way by which plasmatic coagulation starts. TFPI is a potent direct inhibitor of factor Xa and Xa-dependent inhibitor of the VIIa-Tissue Factor (TF) complex. In hemophilic patient, the production of Xa by the amplification pathway being strongly altered because of factor VIII or IX deficiency, thrombin generation (via Xa) comes exclusively from TFPI regulated tissue factor pathway. We can thus say that if haemophilic patients bleed, it is also because of the presence of TFPI that inhibits at the same time Xa and the complex TF-VIIa as soon as factor Xa is generated.

ELIGIBILITY:
Inclusion Criteria:

* Haemophilia A and B patients between 18 and 65 years old, whatever the severity of their disease, who have signed the informed consent form
* On-demand or on prophylactic therapy.
* Regular monitoring in investigator center.

Exclusion Criteria:

* - Haemophilia patients under 18.
* Presence of an inhibitor at any time before or during the study period.
* Patients who received factor VIII concentrate less than 72 hours or factor IX concentrate less than 96 hours before blood collection
* Patients who refused to sign informed consent
* Patient data over the last 5 years at least not available.
* No regular monitoring in haemophilia center (required at least one visit every 18 months for severe or moderate hemophiliac patients).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Haemophilia A and B patients between 18 and 65 years old, whatever the severity of their disease
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2012-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Comparison for TFPI level between Haemophilia A and Haemophilia B | day 1
  Comparison for TFPI level between Haemophilia A and Haemophilia B
Comparison for TFPI level between severe Haemophilia A and severe Haemophilia B | Day 1
  Comparison for TFPI level between severe Haemophilia A and severe Haemophilia B
Comparison for TFPI level between moderate or mild Haemophilia A and moderate or mild Haemophilia B | Day 1
  Comparison for TFPI level between moderate or mild Haemophilia A and moderate or mild Haemophilia B

SECONDARY OUTCOMES:
Correlation between free TFPI and hemorrhagic score | day 1
  Hemorrhagic score is established on the 5 to 10 last years. For severe hemophilic patients: it will use a composite scoring system designed to reflect the clinical severity of haemophilia and named HSS for Haemophilia Severity Score (HSS). It consists in the sum of three components: annual incidence of joint bleeds, orthopedic joint score and annual factor utilization. The orthopedic joint score combines pain and physical examination scores as recommended by the orthopedic Advisory Committee of the World Federation of Haemophilia.
  For mild or moderate hemophilic patients, HSS is not suitable. A composite measure will be used and consist in all bleeding events and consumption of factor concentrate in surgical situation.
  Free TFPI levels will be measured by ELISA according to the manufacturer's recommendations
Correlation between TFPI activity and hemorrhagic score | day 1
  Hemorrhagic score is established on the 5 to 10 last years. For severe hemophilic patients: it will use a composite scoring system designed to reflect the clinical severity of haemophilia and named HSS for Haemophilia Severity Score. It consists in the sum of three components: annual incidence of joint bleeds, orthopedic joint score and annual factor utilization. The orthopedic joint score combines pain and physical examination scores as recommended by the orthopedic Advisory Committee of the World Federation of Haemophilia.
  For mild or moderate hemophilic patients, HSS is not suitable. A composite measure will be used and consist in all bleeding events and consumption of factor concentrate in surgical situation.
  TFPI activity will be measured according to the technique described and modified by Sandset
Correlation between Endogenous Thrombin Potential (ETP) and free TFPI | day 1
  Endogenous Thrombin Potential (i.e. the aera under the thrombin generation curve, nM.min) is measured by thromboplastin Generation Test (TGTs) Free TFPI levels will be measured by ELISA according to the manufacturer's recommendations
Correlation between Lag Time and free TFPI | day 1
  Lag time (min) of the thrombin Generation curve is measured by thromboplastin Generation Test (TGTs) Free TFPI levels will be measured by ELISA according to the manufacturer's recommendations
Correlation between Peak value and free TFPI | day 1
  Peak Value (PV, nmol thrombin) of the thrombin Generation curve is measured by thromboplastin Generation Test (TGTs) Free TFPI levels will be measured by ELISA according to the manufacturer's recommendations
Correlation between Time to Peak and free TFPI | day 1
  Time to Peak (TTP, min) of the thrombin Generation curve is measured by thromboplastin Generation Test (TGTs) Free TFPI levels will be measured by ELISA according to the manufacturer's recommendations
Correlation between ETP and hemorrhagic score | day 1
  Endogenous Thrombin Potential (i.e. the aera under the thrombin generation curve, nM.min) is measured by Thromboplastin Generation Test (TGTs) Hemorrhagic score is established on the 5 to 10 last years. For severe hemophilic patients: it will use a composite scoring system designed to reflect the clinical severity of haemophilia and named HSS for Haemophilia Severity Score. It consists in the sum of three components: annual incidence of joint bleeds, orthopedic joint score and annual factor utilization. The orthopedic joint score combines pain and physical examination scores as recommended by the orthopedic Advisory Committee of the World Federation of Haemophilia.
  For mild or moderate hemophilic patients, HSS is not suitable. A composite measure will be used and consist in all bleeding events and consumption of factor concentrate in surgical situation.
Correlation between Lag Time and hemorrhagic score | day 1
  Lag time (min) of the thrombin generation curve is measured by thromboplastin Generation Test (TGTs) Hemorrhagic score is established on the 5 to 10 last years. For severe hemophilic patients: it will use a composite scoring system designed to reflect the clinical severity of haemophilia and named HSS for Haemophilia Severity Score. It consists in the sum of three components: annual incidence of joint bleeds, orthopedic joint score and annual factor utilization. The orthopedic joint score combines pain and physical examination scores as recommended by the orthopedic Advisory Committee of the World Federation of Haemophilia.
  For mild or moderate hemophilic patients, HSS is not suitable. A composite measure will be used and consist in all bleeding events and consumption of factor concentrate in surgical situation.
Correlation between Peak Value and hemorrhagic score | day 1
  Peak Value (PV, nmol thrombin) of the thrombin generation curve is measured by thromboplastin Generation Test (TGTs) Hemorrhagic score is established on the 5 to 10 last years. For severe hemophilic patients: it will use a composite scoring system designed to reflect the clinical severity of haemophilia and named HSS for Haemophilia Severity Score. It consists in the sum of three components: annual incidence of joint bleeds, orthopedic joint score and annual factor utilization. The orthopedic joint score combines pain and physical examination scores as recommended by the orthopedic Advisory Committee of the World Federation of Haemophilia.
  For mild or moderate hemophilic patients, HSS is not suitable. A composite measure will be used and consist in all bleeding events and consumption of factor concentrate in surgical situation.
Correlation between Time to Peak and hemorrhagic score | day 1
  Time to Peak (TTP, min) of the thrombin generation curve is measured by thromboplastin Generation Test (TGTs) Hemorrhagic score is established on the 5 to 10 last years. For severe hemophilic patients: it will use a composite scoring system designed to reflect the clinical severity of haemophilia and named HSS for Haemophilia Severity Score. It consists in the sum of three components: annual incidence of joint bleeds, orthopedic joint score and annual factor utilization. The orthopedic joint score combines pain and physical examination scores as recommended by the orthopedic Advisory Committee of the World Federation of Haemophilia.
  For mild or moderate hemophilic patients, HSS is not suitable. A composite measure will be used and consist in all bleeding events and consumption of factor concentrate in surgical situation.
Comparison for ETP between haemophilia A et Haemophilia B | Day 1
  Endogenous Thrombin Potential (i.e. the aera under the thrombin generation curve, nM.min) is measured by Thromboplastin Generation Test (TGTs)
Comparison for lag time between haemophilia A et Haemophilia B | Day 1
  Lag time (min) of the thrombin generation curve is measured by thromboplastin Generation Test (TGTs)
Comparison for Peak Value between haemophilia A et Haemophilia B | Day 1
  Peak Value (PV, nmol thrombin) of the thrombin generation curve is measured by thromboplastin Generation Test (TGTs)
Comparison for Time to Peak between haemophilia A et Haemophilia B | day 1
  Time to Peak (TTP, min) of the thrombin generation curve is measured by thromboplastin Generation Test (TGTs)

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHRU Lille, Lille
  - HCL, Lyon
  - AP-HM, Marseille
  - Chu Nancy, Nancy
  - Chu Reims, Reims
  - CHU Saint-Etienne, Saint-Etienne
  - Chu Tours, Tours